CLINICAL TRIAL: NCT06268925
Title: The Feasibility And Efficacy Of A Telerehabilitation Program For People With Knee Osteoarthiritis In Sri Lanka
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: University of Peradeniya (Other)
Responsible Party: Principal Investigator, M.S.F.Sarjana, Principal investigator, University of Peradeniya
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: UAHS
Record Dates: First submitted 2023-12-02; First posted 2024-02-20 (Actual); Last update posted 2024-02-20 (Actual); Status verified 2024-02

CONDITIONS: Knee Osteoarthritis
Keywords: Telerehabilitation; Feasibility; Efficacy; Sri Lanka
MeSH Terms: conditions — Osteoarthritis, Knee | interventions — Exercise

STUDY DESIGN:
Intervention Model Description: 14 people with knee osteoarthritis will be recruited and conducted group classes through zoom
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Study group (Experimental): single arm group exercises will be given to the patients
  Interventions: Other: Exercises

INTERVENTIONS:
Other: Exercises — number of exercises will be guided to do through zoom

SUMMARY:
it will be 8 week zoom program of exercises for knee osteo arthritis. participant will be selected according to elegibilty criteria. pre and post measurements will be obtained. then feasibility and efficacy will be assesed.

DETAILED DESCRIPTION:
This research is to check the feasibility and efficacy of a telerehabilitation program for people with knee osteoarthritis in Sri Lanka. 14 people with knee OA will be recruited according to the inclusion and exclusion criteria. Study group will be selected with advertisement on facebook.

People who are interested will be included. Exercise booklet and instruction materials will be given to patients and initial measurement of Pain using VAS scale, 30 CST (30 second chair stand test)- Lower extremity muscle strength and dynamic balance, WOMAC (Western Ontario and McMaster Universities Arthritis Index)- pain, stiffness and physical activity will be obtained. Study group will go for 8 weeks of zoom program of exercises. Classes will be taken by the physiotherapist 3 days per week with standardized program called PEAK.knee log book will be maintained by therapist. Post 8 week same measurements on baseline will be reassessed and additional to that, Feasibility and acceptability for tele rehabilitation and Patient adherence and Safety will be assessed with attrition rate, satisfaction rate , participation to the program and measuring adverse effect respectively. Statistical Package for Social Science (SPSS) version for Windows will be used for data analysis. Pair t test will be used to compare the baseline and post 8 week results.

ELIGIBILITY:
Inclusion Criteria:

Meet National Institute for Health and Care Excellence clinical criteria for OA

* Age ≥45 years.
* Activity-related knee joint pain.
* Morning knee stiffness ≤ 30 min.
* Report history of knee pain ≥ 3mths.
* Report knee pain on most days of the past month.
* Report an average pain score of at least 4 on an 11-point numeric rating scale during walking over the previous week.
* Report difficulty walking and climbing stairs.
* Have access to a device with internet connection: if they can use without assistance if possible

Exclusion Criteria:

* On waiting list for/planning knee/hip surgery in next 12 months.
* Previous arthroplasty on affected knee.
* Recent knee surgery (past 6 months).
* Consulting/ed physiotherapy or doing strengthening exercise for knee (past 6 months).
* Self-reported inflammatory arthritis (eg rheumatoid arthritis).
* Any neurological condition affecting lower limbs; and/or any unstable/uncontrolled cardiovascular condition.
* Clearance to participate from a general practitioner will be required for anyone who reported a fall (past 12 months) or is house-bound due to immobility

Min Age: 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 14 (Estimated)
Dates: Start 2024-02-22 (Estimated); Primary Completion 2024-04-22 (Estimated); Study Completion 2024-05-03 (Estimated)

PRIMARY OUTCOMES:
Efficacy of telerehabilitation program | post 8 weeks of exercise program
  measured by attrition rate which is the measure of screened individual who are eligible but refused to participate and proportion of screened individuals who enrolled in to the study
Feasibility and acceptability | post 8 week
  asking patients "how satisfied they are about tele rehabilitation program" respectively at 8 weeks post.

SECONDARY OUTCOMES:
lower extremity muscle strength and dynamic balance | pre and post 8 week of exercise program
  30 second chair stand test
pain, | Pre and post 8 weeks of exercise program
  assessed by Visual Analogue Scale containing 0 to 10 scale
pain stiffness and physical activity | pre and post 8 week of exercise program
  WOMAC scale (Western Ontario and McMaster Universities Arthritis Index)

CONTACTS AND LOCATIONS:
Locations (1):
- M.S.F.Sarjana, Puttalam, North Western Province, Sri Lanka

IPD SHARING:
Plan to Share IPD: No